CLINICAL TRIAL: NCT04238104
Title: Study on the Normal Range of Pulse Oximetry and the Threshold for Screening Critical Congenital Heart Disease in Neonates at Different Altitudes in China
Brief Title: POX Range and the Threshold for Screening Major CHD in Neonates at Different Altitudes
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Hainan women and children medical center (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Qinghai Red Cross Hospital (Other); Tibet Autonomous Region People's Hospital (Other); People's Hospital of Golog Tibetan Autonomous Prefecture (Unknown); People's Hospital of Naqu District, Tibet (Unknown); People's Hospital of Luchun County, Yunnan Province (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-296
Record Dates: First submitted 2019-11-26; First posted 2020-01-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-12

CONDITIONS: POX Range of Healthy Newborns at Different Altitudes; POX Threshold for Screening Major CHD in Neonates
Keywords: Saturation; Cut-off value; Neonates; Altitude; POX; major CHD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- sea level: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center of sea level were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention
- altitude <1000: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center with the altitude less than 1000 metres were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention
- altitude 1000-2000: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center with the altitude between 1000-2000 metres were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention
- altitude 2000-3000: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center with the altitude between 2000-3000 metres were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention
- altitude 3000-4000: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center with the altitude between 3000-4000 metres were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention
- altitude 4000-5000: Pulse oximetry was performed between 6 and 72 hours after delivery (measured and recorded at 6, 12, 24, 48 and 72 hours respectively). Using Masimo Radical-7 (Irvine, CA, USA) to measure. All measurements at the medical center with the altitude between 4000-5000 metres were performed by the well-trained investigator. All major CHD infants will be measured the POX by the same way during the whole study period.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — it's only observational study. No interventions.

SUMMARY:
major CHD (Congenital Heart Disease) screening by POX (pulse oximetry) in sea-level areas is not fit for low, medium and high altitude areas, but the normal range of pulse oximetry at different altitude areas has not been studied before, so the current screening technology can only be used in sea-level areas, but not for newborns in low, medium and high altitude areas. We need to carry out a research to clarify the range of POX and make sure the threshold of POX in major CHD screening in different altitude areas of China.

DETAILED DESCRIPTION:
At present, the application of POX (pulse oximetry) in screening major CHD (congenital heart disease ) has been legislated in the United States. In China, the two indicators of POX plus auscultation of heart murmur for screening major CHD have also been promoted as national standards. There are differences in the POX range of newborns at different altitude areas, so the threshold of POX screening based on sea-level areas is not applicable to low, medium and high altitude areas. While the normal range of POX at different altitude areas has not been studied in detail, so the current screening strategy can only be used in sea-level areas, but not benefit newborns in low, medium and high altitude areas. In order to apply major CHD screening strategy better to cover the newborns all over the country, we need to clarify the range of POX at different altitude areas of China and make sure the threshold of POX in major CHD screening. We plan to carry out a multicenter study on the normal POX value range of healthy and asymptomatic term newborns 6-72 hours after delivery in medical centers with altitude of 500-1000; 1000-2000; 2000-3000; 3000-4000 and above 4000 meters. And compare the POX value at different altitude areas with that of newborns delivered in the maternity hospitals at sea level. And measure the POX value of newborns with major CHD in the same way. POX screening thresholds will be obtained at different altitude areas. We will test the hypothesis that POX of healthy newborns at different altitude areas is lower than that of healthy newborns at sea level, and POX threshold of major CHD screening is lower than that of sea level.

ELIGIBILITY:
Inclusion Criteria:

For healthy newborns:

* Healthy, asymptomatic, singleton term infants (37-41 weeks gestation);
* Appropriate for gestational age (using the international WHO's intrauterine growth curve to evaluate);
* Only newborns with Apgar score ≥ 7 in 1 minute and 5 minutes were selected;
* There is no known congenital heart disease based on the ECHO result , no murmur, no obvious signs (no fever, no tachycardia or respiratory symptoms at the time of admission).

For major CHD newborns:

* Echocardiography clearly diagnosed the following congenital heart diseases: Aortic stenosis, Double outlet of right ventricle, Ebstein's malformation, Left cardiac hypoplasia syndrome, Aortic arch disconnection, Pulmonary atresia, Single ventricle, Tetralogy of Fallot, Complete anomalous pulmonary venous drainage, Transposition of great arteries, Tricuspid valve atresia, and Single trunk of arteries and other major CHD based on Ewer's denition.

Exclusion Criteria:

For healthy newborns:

* Newborn with caesarean section; newborn with smoking mother; newborn with definite congenital heart disease before discharge.

For major CHD newborns:

* There is no exclusion criteria for major CHD.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: During the study period (January 15, 2019 to December 15, 2020), all newborns in continuous delivery were included simultaneously in various medical centers in different altitude areas. For major CHD infants, the study period will be January 15, 2019 to December 15, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Pulse oximetry of healthy newborns at 6th hour after birth at different altitudes | At 6th hours after birth
  Pulse oximetry of healthy newborns at 6th hour after birth would be measured by monitor at 6th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.

SECONDARY OUTCOMES:
Pulse oximetry of healthy newborns at 12th hour after birth at different altitudes | At 12th hours after birth
  Pulse oximetry of healthy newborns at 12th hour after birth would be measured by monitor at 12th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of healthy newborns at 24th hour after birth at different altitudes | At 24th hours after birth
  Pulse oximetry of healthy newborns at 24th hour after birth would be measured by monitor at 24th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of healthy newborns at 48th hour after birth at different altitudes | At 48th hours after birth
  Pulse oximetry of healthy newborns at 48th hour after birth would be measured by monitor at 48th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of healthy newborns at 72th hour after birth at different altitudes | At 72th hours after birth
  Pulse oximetry of healthy newborns at 72th hour after birth would be measured by monitor at 72th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of newborns with critical congenital heart disease at 6th hour after birth at different altitudes | At 6th hours after birth
  Pulse oximetry of critical congenital heart disease newborns at 6th hour after birth would be measured by monitor at 6th hour after birth and would be described by range interquartile in critical congenital heart disease neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of newborns with critical congenital heart disease at 12th hour after birth at different altitudes | At 12th hours after birth
  Pulse oximetry of critical congenital heart disease newborns at 12th hour after birth would be measured by monitor at 12th hour after birth and would be described by range interquartile in healthy neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of newborns with critical congenital heart disease at 24th hour after birth at different altitudes | At 24th hours after birth
  Pulse oximetry of critical congenital heart disease newborns at 24th hour after birth would be measured by monitor at 24th hour after birth and would be described by range interquartile in critical congenital heart disease neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of newborns with critical congenital heart disease at 48th hour after birth at different altitudes | At 48th hours after birth
  Pulse oximetry of critical congenital heart disease newborns at 48th hour after birth would be measured by monitor at 48th hour after birth and would be described by range interquartile in critical congenital heart disease neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.
Pulse oximetry of newborns with critical congenital heart disease at 72th hour after birth at different altitudes | At 72th hours after birth
  Pulse oximetry of critical congenital heart disease newborns at 72th hour after birth would be measured by monitor at 72th hour after birth and would be described by range interquartile in critical congenital heart disease neonates in hospitals with different altitudes.
  Altitude levels :sea level, within 1000 meters above sea level, 1000 to 2000 meters above sea level, 2000 to 3000 meters above sea level, 3000 to 4000 meters above sea level and 4000 to 5000 meters above sea level.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Yan, PhD, Study Chair — Epidemiology Office of Children's hospital of Fudan University
Locations (8):
- China (8):
  - People's Hospital of Golog Tibetan Autonomous Prefecture, Guoluo Prefecture
  - Hainan women and children medical center, Haikou
  - Yan'an Hospital Affiliated to Kunming Medical University, Kunming
  - Tibet Autonomous People's Hospital, Lhasa
  - People's Hospital of Luchun County, Yunnan Province, Luchun
  - People's Hospital of Naqu District, Tibet, Naqu
  - Qinghai Red Cross Hospital, Qinghai
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi

IPD SHARING:
Plan to Share IPD: No